CLINICAL TRIAL: NCT04545333
Title: Real World Observational Study Using clonoSEQ® Next Generation Sequencing in Hematologic Malignancies: The 'Watch' Registry
Brief Title: The clonoSEQ® Watch Registry
Status: Terminated | Type: Observational
Why Stopped: Sufficient data collected.
Sponsor: Adaptive Biotechnologies (Industry)
Responsible Party: Sponsor
Other Study IDs: ADAP-008
Record Dates: First submitted 2020-08-31; First posted 2020-09-11 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Acute Lymphoblastic Leukemia, Adult B-Cell; Chronic Lymphocytic Leukemia; Multiple Myeloma; Non-hodgkin Lymphoma
Keywords: Minimal residual disease; measurable residual disease; MRD; clonoSEQ; ALL; CLL; MM; NHL; Watch Registry
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Lymphoma, Non-Hodgkin; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Remaining samples will be stored for potential use in future assay development research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- ALL: patients diagnosed with acute lymphoblastic leukemia
  Interventions: Diagnostic Test: clonoSEQ Assay
- CLL: patients diagnosed with chronic lymphocytic leukemia
  Interventions: Diagnostic Test: clonoSEQ Assay
- MM: patients diagnosed with multiple myeloma
  Interventions: Diagnostic Test: clonoSEQ Assay
- NHL: patients diagnosed with non-Hodgkin lymphoma
  Interventions: Diagnostic Test: clonoSEQ Assay

INTERVENTIONS:
Diagnostic Test: clonoSEQ Assay — minimal residual disease (MRD) assay using blood, bone marrow, or other tissue containing tumor cells

SUMMARY:
This is a prospective, multicenter, observational study of adult patients with a diagnosis of acute lymphoblastic leukemia (ALL), multiple myeloma (MM), chronic lymphocytic leukemia (CLL), or non-Hodgkin lymphoma (NHL). This study will enroll up to 528 patients in up to 50 sites in the United States and collect data with regard to use of the clonoSEQ MRD assay in the management of lymphoid malignancies.

DETAILED DESCRIPTION:
Data show that detection of MRD may be important to guide treatment decisions in ALL, MM, CLL, and NHL. However, there remains a lack of real-world evidence for making therapeutic decisions based upon MRD status. This study is designed to understand when in a patient's treatment continuum the assay is used and how clonoSEQ MRD data impact the treatment decisions made by investigators.

All patients enrolled in the study will be followed for at least 2 yrs. Demographic data and disease status will be captured at study enrollment. Patients must be >/= 18 yrs of age and able to sign informed consent. A given patient is eligible to enroll in the study if the treating physician has made the decision to use the clonoSEQ assay as part of that patient's routine cancer care. Reasons for placing a clonoSEQ order and subsequent decisions made as a result of MRD data will be tracked. Patient treatment will also be tracked over the course of the study in order to understand how clonoSEQ use is incorporated into current treatment regimens.

Participating centers will include sites that actively use clonoSEQ to manage their patients with lymphoid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to provide written informed consent
2. A decision has been made by the treating provider to use the clonoSEQ Assay as part of routine clinical care
3. Age ≥ 18 years;
4. Documented hematologic malignancy (any of the below):

   1. MM
   2. ALL (B and T-cell subtypes)
   3. B-cell NHL (all sub types)
   4. CLL
   5. Other lymphoid malignancies (upon review and approval by study chair)

Exclusion Criteria:

Patients must not meet any of the following criteria in order to be enrolled into the study:

1. Concurrent enrollment in a clinical trial where treatment decisions and patterns are dictated per protocol
2. A decision has been made by the treating provider to not use the clonoSEQ Assay as part of routine clinical care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of ALL, MM, CLL, or NHL whose SOC response assessments will include monitoring of MRD status by clonoSEQ Assay
Sampling Method: Non-Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Distribution of timepoints at which MRD is monitored using the clonoSEQ Assay in lymphoid malignancy patients in real world settings | up to 3 yrs
  Data will be collected to determine at what points lymphoid malignancy patients are in their treatment continuums when the clonoSEQ Assay is used to monitor MRD levels

SECONDARY OUTCOMES:
Numbers of lymphoid malignancy patients with intensifications to their drug regimens based upon clonoSEQ MRD results | up to 3 yrs
  Data will be collected with regard to changes to treatment/drug regimens in order to determine how clonoSEQ Assay MRD results inform and impact routine clinical practice
Numbers of lymphoid malignancy patients with de-intensifications to their drug regimens based upon clonoSEQ MRD results | up to 3 yrs
  Data will be collected with regard to changes to treatment/drug regimens in order to determine how clonoSEQ Assay MRD results inform and impact routine clinical practice

OTHER OUTCOMES:
Average numbers of clonoSEQ Assay orders placed for enrolled lymphoid malignancy patients in routine clinical practice relative to other response assessments | up to 3 yrs
  Data will be collected to determine how the clonoSEQ Assay is used as part of routine disease response assessments in lymphoid malignancy patients
Differences in outcomes between clonoSEQ Assay MRD-negative and MRD-positive lymphoid malignancy patients | up to 3 yrs
  Data will be collected to assess the following, as applicable, depending upon distribution of patients that enroll in this study:
  * Response to treatment, duration of response, time to next therapy, duration of maintenance therapy, and survival
  * Numbers of patients who proceed to transplant in the ALL and MM cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Simmons, PhD, Study Director — Adaptive Biotechnologies
Locations (14):
- United States (14):
  - Stanford Hospital, Stanford, California
  - Georgetown University, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Edward H. Kaplan MD & Associates, Skokie, Illinois
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - American Oncology Partners of Maryland, Bethesda, Maryland
  - Washington University, St Louis, Missouri
  - Novant Health, Charlotte, North Carolina
  - Oregon Health & Science University, Knight Cancer Institute, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Bon Secours St Francis, Greenville, South Carolina
  - University of Washington, Seattle Cancer Care Alliance, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Undecided